CLINICAL TRIAL: NCT02246361
Title: Impact of Six Patient Information Leaflets (PIL) on Doctor Patient Communication and Adherence in Emergency Ward
Brief Title: Impact of Six Patient Information Leaflets (PIL) on Doctor Patient Communication
Acronym: EDIFIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Floralis (Industry)
Collaborators: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N°IRB 5891
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Ankle Sprain; Infectious Colitis; Diverticulitis; Pyelonephritis; Prostatitis; Pneumonitis
Keywords: Ankle sprain; Infectious colitis; Diverticulitis; Pyelonephritis; Prostatitis; Pneumonitis; Patient Information Leaflet (PIL); Doctor Patient Communication; Adherence; Satisfaction; Scale; Doctor Patient Communication scale; Adherence scale; Satisfaction scale
MeSH Terms: conditions — Ankle Injuries; Diverticulitis; Pyelonephritis; Prostatitis; Pneumonia; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 (without PIL) (No Intervention): No particular intervention during consultation for the patient
- Phase 2 (Experimental): Patient Information Leaflet is given to the patient during the consultation
  Interventions: Procedure: Patient Information Leaflet (PIL)

INTERVENTIONS:
Procedure: Patient Information Leaflet (PIL) — Patient Information Leaflet (PIL) about infectious colitis, diverticulitis, pneumonitis, prostatitis or either pyelonephritis is given to the patient related to his disease during the consultation
  Arms: Phase 2

SUMMARY:
The purpose of this "before-after" prospective multicenter study is to assess the impact of six Patient Information Leaflets (PILs) on Doctor Patient Communication scale (DPC) and adherence scale for common acute illnesses in emergency ward.

DETAILED DESCRIPTION:
Assessing the impact of six Patient Information Leaflets (PILs) on Doctor Patient Communication scale (DPC) and adherence scale for common acute illnesses (infectious colitis, diverticulitis, pneumonitis, prostatitis, pyelonephritis , ankle sprain) in two emergency ward.

For "before" study without intervention : usual consultation without PIL .

For "after study" with intervention : the patient is given a PIL related to his disease during the consultation.

Data collection will take place the same day as the consultation by self-administered questionnaire for DPC scale and also between 7 to 10 days after the consultation by phone survey for DPC scale and adherence scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient.
* Minor aged over 15 years accompanied by a responsible adult.
* The patient must be reachable by telephone within seven to ten days following the consultation.

Exclusion Criteria:

* Illiterate patient.
* Patient refusing follow-up call.
* Patient with visual or hearing impairment.
* Patient non-Francophone.
* Private patient of liberty by judicial or administrative.
* Person being a measure of legal protection.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Doctor Patient Communication score | In seven to ten days after delivery
  All patients will be called seven to ten days after the delivery of a PIL during the visit to answer a questionnaire on their perception of Doctor Patient Communication (DPC) since they visit the GP. Il will permit to calculate a DPC score.

SECONDARY OUTCOMES:
Adherence score | In seven to ten days after the delivery
  All patients will be called seven to ten days after the delivery of a PIL during the visit, to answer a questionnaire on their adherence related to the disease since they visit the GP. Il will permit to calculate a adherence score.
Satisfaction score | In seven to ten days after the delivery
  All patients will be called seven to ten days after the visit, to answer a questionnaire on their satisfaction about since they visit the GP. Il will permit to calculate a satisfaction score.
Doctor Patient Communication score | Just after the visit
  All patients will answer to a self questionnaire on their perception of Doctor Patient Communication (DPC) just after the visit of the GP. Il will permit to calculate a DPC score.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Sustersic, MD, Principal Investigator — Floralis France
Locations (2):
- France (2):
  - Groupe Hospitalier Mutualiste, service des urgences, Grenoble, Isere
  - Centre Hospitalier, Chambéry, Savoie

REFERENCES:
- [Background] Sustersic M, Jeannet E, Cozon-Rein L, Marechaux F, Genty C, Foote A, David-Tchouda S, Martinez L, Bosson JL. Impact of information leaflets on behavior of patients with gastroenteritis or tonsillitis: a cluster randomized trial in French primary care. J Gen Intern Med. 2013 Jan;28(1):25-31. doi: 10.1007/s11606-012-2164-8. Epub 2012 Jul 25. PMID 22829293
- [Background] Sustersic M, Meneau A, Dremont R, Paris A, Laborde L, Bosson JL. [Developing patient information sheets in general practice. Proposal for a methodology]. Rev Prat. 2008 Dec 15;58(19 Suppl):17-24. French. PMID 19253787
- [Background] Little P, Moore M, Kelly J, Williamson I, Leydon G, McDermott L, Mullee M, Stuart B; PIPS Investigators. Delayed antibiotic prescribing strategies for respiratory tract infections in primary care: pragmatic, factorial, randomised controlled trial. BMJ. 2014 Mar 6;348:g1606. doi: 10.1136/bmj.g1606. PMID 24603565
- [Background] Coudeyre E, Tubach F, Rannou F, Baron G, Coriat F, Brin S, Revel M, Poiraudeau S. Effect of a simple information booklet on pain persistence after an acute episode of low back pain: a non-randomized trial in a primary care setting. PLoS One. 2007 Aug 8;2(8):e706. doi: 10.1371/journal.pone.0000706. PMID 17684553
- [Background] Grime J, Blenkinsopp A, Raynor DK, Pollock K, Knapp P. The role and value of written information for patients about individual medicines: a systematic review. Health Expect. 2007 Sep;10(3):286-98. doi: 10.1111/j.1369-7625.2007.00454.x. PMID 17678517
- [Background] Gauchet A, Tarquinio C, Fischer G. Psychosocial predictors of medication adherence among persons living with HIV. Int J Behav Med. 2007;14(3):141-50. doi: 10.1007/BF03000185. PMID 18062057
- [Background] Nicolson D, Knapp P, Raynor DK, Spoor P. Written information about individual medicines for consumers. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD002104. doi: 10.1002/14651858.CD002104.pub3. PMID 19370575
- [Background] Fox R. Informed choice in screening programmes: do leaflets help? A critical literature review. J Public Health (Oxf). 2006 Dec;28(4):309-17. doi: 10.1093/pubmed/fdl066. Epub 2006 Oct 23. PMID 17060352
- [Background] Graham W, Smith P, Kamal A, Fitzmaurice A, Smith N, Hamilton N. Randomised controlled trial comparing effectiveness of touch screen system with leaflet for providing women with information on prenatal tests. BMJ. 2000 Jan 15;320(7228):155-60. doi: 10.1136/bmj.320.7228.155. PMID 10634736
- [Background] Kenny T, Wilson RG, Purves IN, Clark J Sr, Newton LD, Newton DP, Moseley DV. A PIL for every ill? Patient information leaflets (PILs): a review of past, present and future use. Fam Pract. 1998 Oct;15(5):471-9. doi: 10.1093/fampra/15.5.471. PMID 9848435
- [Background] Little P, Dorward M, Warner G, Moore M, Stephens K, Senior J, Kendrick T. Randomised controlled trial of effect of leaflets to empower patients in consultations in primary care. BMJ. 2004 Feb 21;328(7437):441. doi: 10.1136/bmj.37999.716157.44. Epub 2004 Feb 13. PMID 14966078
- [Background] Raynor DK, Blenkinsopp A, Knapp P, Grime J, Nicolson DJ, Pollock K, Dorer G, Gilbody S, Dickinson D, Maule AJ, Spoor P. A systematic review of quantitative and qualitative research on the role and effectiveness of written information available to patients about individual medicines. Health Technol Assess. 2007 Feb;11(5):iii, 1-160. doi: 10.3310/hta11050. PMID 17280623
- [Background] Paris A, Cornu C, Auquier P, Maison P, Radauceanu A, Brandt C, Salvat-Melis M, Hommel M, Cracowski JL. French adaptation and preliminary validation of a questionnaire to evaluate understanding of informed consent documents in phase I biomedical research. Fundam Clin Pharmacol. 2006 Feb;20(1):97-104. doi: 10.1111/j.1472-8206.2005.00391.x. PMID 16448400
- [Background] Zapata LB, Steenland MW, Brahmi D, Marchbanks PA, Curtis KM. Patient understanding of oral contraceptive pill instructions related to missed pills: a systematic review. Contraception. 2013 May;87(5):674-84. doi: 10.1016/j.contraception.2012.08.026. Epub 2012 Oct 4. PMID 23040136
- [Background] Ziegler A, Hadlak A, Mehlbeer S, Konig IR. Comprehension of the description of side effects in drug information leaflets: a survey of doctors, pharmacists and lawyers. Dtsch Arztebl Int. 2013 Oct;110(40):669-73. doi: 10.3238/arztebl.2013.0669. Epub 2013 Oct 4. PMID 24167524
- [Background] Talen MR, Muller-Held CF, Eshleman KG, Stephens L. Patients' communication with doctors: a randomized control study of a brief patient communication intervention. Fam Syst Health. 2011 Sep;29(3):171-83. doi: 10.1037/a0024399. PMID 21787080
- [Background] Macfarlane J, Holmes W, Gard P, Thornhill D, Macfarlane R, Hubbard R. Reducing antibiotic use for acute bronchitis in primary care: blinded, randomised controlled trial of patient information leaflet. BMJ. 2002 Jan 12;324(7329):91-4. doi: 10.1136/bmj.324.7329.91. PMID 11786454
- [Background] Francis NA, Butler CC, Hood K, Simpson S, Wood F, Nuttall J. Effect of using an interactive booklet about childhood respiratory tract infections in primary care consultations on reconsulting and antibiotic prescribing: a cluster randomised controlled trial. BMJ. 2009 Jul 29;339:b2885. doi: 10.1136/bmj.b2885. PMID 19640941
- [Background] Johnson A, Sandford J. Written and verbal information versus verbal information only for patients being discharged from acute hospital settings to home: systematic review. Health Educ Res. 2005 Aug;20(4):423-9. doi: 10.1093/her/cyg141. Epub 2004 Nov 30. PMID 15572437
- [Background] Johnson A, Sandford J, Tyndall J. Written and verbal information versus verbal information only for patients being discharged from acute hospital settings to home. Cochrane Database Syst Rev. 2003;2003(4):CD003716. doi: 10.1002/14651858.CD003716. PMID 14583990
- [Background] Little P, Rumsby K, Kelly J, Watson L, Moore M, Warner G, Fahey T, Williamson I. Information leaflet and antibiotic prescribing strategies for acute lower respiratory tract infection: a randomized controlled trial. JAMA. 2005 Jun 22;293(24):3029-35. doi: 10.1001/jama.293.24.3029. PMID 15972565
- [Background] Allenet B, Baudrant M, Lehmann A, Gauchet A, Roustit M, Bedouch P, Golay A. [How can we evaluate medication adherence? What are the methods?]. Ann Pharm Fr. 2013 Mar;71(2):135-41. doi: 10.1016/j.pharma.2012.10.001. Epub 2012 Nov 6. French. PMID 23537415
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Wells FO. Patient information--the present and the future. J R Soc Med. 1990 May;83(5):300-2. doi: 10.1177/014107689008300507. No abstract available. PMID 2380945
- [Background] Finnie RK, Felder TM, Linder SK, Mullen PD. Beyond reading level: a systematic review of the suitability of cancer education print and Web-based materials. J Cancer Educ. 2010 Dec;25(4):497-505. doi: 10.1007/s13187-010-0075-0. PMID 20237884
- [Background] Carre PC, Roche N, Neukirch F, Radeau T, Perez T, Terrioux P, Ostinelli J, Pouchain D, Huchon G. The effect of an information leaflet upon knowledge and awareness of COPD in potential sufferers. A randomized controlled study. Respiration. 2008;76(1):53-60. doi: 10.1159/000115947. Epub 2008 Feb 5. PMID 18253024
- [Background] Heaney D, Wyke S, Wilson P, Elton R, Rutledge P. Assessment of impact of information booklets on use of healthcare services: randomised controlled trial. BMJ. 2001 May 19;322(7296):1218-21. doi: 10.1136/bmj.322.7296.1218. PMID 11358776
- [Background] Yardley L, Barker F, Muller I, Turner D, Kirby S, Mullee M, Morris A, Little P. Clinical and cost effectiveness of booklet based vestibular rehabilitation for chronic dizziness in primary care: single blind, parallel group, pragmatic, randomised controlled trial. BMJ. 2012 Jun 6;344:e2237. doi: 10.1136/bmj.e2237. PMID 22674920
- [Background] Smith SK, Trevena L, Simpson JM, Barratt A, Nutbeam D, McCaffery KJ. A decision aid to support informed choices about bowel cancer screening among adults with low education: randomised controlled trial. BMJ. 2010 Oct 26;341:c5370. doi: 10.1136/bmj.c5370. PMID 20978060
- [Background] Turpin G, Downs M, Mason S. Effectiveness of providing self-help information following acute traumatic injury: randomised controlled trial. Br J Psychiatry. 2005 Jul;187:76-82. doi: 10.1192/bjp.187.1.76. PMID 15994575
- [Background] Cunningham JA, Neighbors C, Wild C, Humphreys K. Ultra-brief intervention for problem drinkers: results from a randomized controlled trial. PLoS One. 2012;7(10):e48003. doi: 10.1371/journal.pone.0048003. Epub 2012 Oct 24. PMID 23110157
- [Background] Felley C, Perneger TV, Goulet I, Rouillard C, Azar-Pey N, Dorta G, Hadengue A, Frossard JL. Combined written and oral information prior to gastrointestinal endoscopy compared with oral information alone: a randomized trial. BMC Gastroenterol. 2008 Jun 3;8:22. doi: 10.1186/1471-230X-8-22. PMID 18522729
- [Background] Galaal K, Bryant A, Deane KH, Al-Khaduri M, Lopes AD. Interventions for reducing anxiety in women undergoing colposcopy. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD006013. doi: 10.1002/14651858.CD006013.pub3. PMID 22161395
- [Derived] Sustersic M, Tissot M, Tyrant J, Gauchet A, Foote A, Vermorel C, Bosson JL. Impact of patient information leaflets on doctor-patient communication in the context of acute conditions: a prospective, controlled, before-after study in two French emergency departments. BMJ Open. 2019 Feb 20;9(2):e024184. doi: 10.1136/bmjopen-2018-024184. PMID 30787085